CLINICAL TRIAL: NCT01503567
Title: Epidemiological Study on Haemophilia Care and Orthopaedic Status in Developing Countries
Acronym: HAEMOcare
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-3971; U1111-1124-6665 (Other: WHO)
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia A With Inhibitors; Haemophilia B; Haemophilia B With Inhibitors
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Subjects 6 to 18 years old without inhibitors
  Interventions: Other: No treatment given
- Subjects 6 to 18 years old with inhibitors
  Interventions: Other: No treatment given
- Subjects above18 years old without inhibitors
  Interventions: Other: No treatment given
- Subjects above 18 years old with inhibitors
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will only fill out a questionaire

SUMMARY:
This study is conducted in Africa and Asia. The aim of this study is to evaluate in the participating countries the orthopaedic status and the degree of arthropathy of severe haemophilia patients in general.

ELIGIBILITY:
Inclusion Criteria:

* Patient (and/or parents or the patient's legally acceptable representative, if applicable) must give signed and dated informed consent before enrolment in the study
* Male patients at least 6 years old with diagnosis of severe congenital haemophilia A or B with or without inhibitors
* Patients receiving on demand replacement factors/bypassing agents therapy

Exclusion Criteria:

* Clinically relevant coagulation disorders other than congenital haemophilia A or B
* Patients on currently active treatment for HCV (Hepatitis C Virus) or HIV (Human Immune Deficiency Virus) infections

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male patients at least 6 years old with severe congenital haemophilia A or B (FVIII or FIX activities below 1% or level below 1U dL^-1) without inhibitor or with inhibitors against FVIII or FIX
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Type of haemophilia and inhibitor characteristics: Against FVIII or FIX; high or low titre; anamnestic response (high or low responder) | After 6 months (recruitment and data collection)
Clinical (using Haemophilia joint score) and radiological (using Pettersson score) orthopaedic status of defined joints: Elbow, knees and ankles in relation to haemophilia A or B | After 6 months (recruitment and data collection)

SECONDARY OUTCOMES:
Mean orthopaedic score in the 4 groups according to the Pettersson and Haemophilia joint scores | After 6 months (recruitment and data collection)
Usage of anti haemophilic treatment in IU/kg | During the last year preceding patient recruitment
Quality of Life - EQ-5D (Euro Quality - 5 Domains) questionnaire | After 6 months (recruitment and data collection)
Economic aspects of the management of haemophiliacs and its burden on patient/family and community resources | After 6 months (recruitment and data collection)
Living characteristics of the patient's household | After 6 months (recruitment and data collection)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Casablanca, Morocco
- Novo Nordisk Investigational Site, Muscat, Oman
- Novo Nordisk Investigational Site, Sandton, South Africa

REFERENCES:
- [Result] Gupta N, Belhani M, Benbouzid A, Andaloussi M El, Maani K, Mahlangu J, Wali Y, Saad HA, Fegoun SB el. The Haemocare Protocol - A composite method to measure the disease burden from Haemophilia in developing countries. European Hematology Association 2013; Country: Sweden City: Stockholm
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com